CLINICAL TRIAL: NCT00366860
Title: Effect of Soy Bread on Markers of Bone Metabolism and Cardiovascular Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Mary A.M. Rogers, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GCRC Protocol #1971
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporosis; Cardiovascular Diseases
Keywords: soy; isoflavones; bone resorption; osteogenesis; diet; hyperlipidemia
MeSH Terms: conditions — Osteoporosis; Cardiovascular Diseases; Bone Resorption; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy bread (Experimental): Soy bread (75-100 mg isoflavone/day) for 12 weeks
  Interventions: Behavioral: Soy bread
- Wheat bread (Active Comparator): Wheat bread for 12 weeks
  Interventions: Behavioral: Soy bread

INTERVENTIONS:
Behavioral: Soy bread

SUMMARY:
A study was designed with two specific aims: (1) to assess the effect of soy bread, compared with wheat bread, on markers of bone metabolism and cardiovascular health, and (2) to evaluate whether soy bread consumption affects the metabolism of phytoestrogens. To answer Aim 1, a double-blind randomized crossover trial was conducted. Individuals with an ability to metabolize a specific isoflavone, daidzein, consumed 3 slices of bread (either soy or wheat) daily over a 12-week period. After a 4-week wash-out period, subjects consumed 3 slices/day of the other type of bread. Markers of bone metabolism and cardiovascular health were evaluated before and after each time period. To answer Aim 2, individuals who did not metabolize daidzein at baseline entered a double-blind randomized trial of soy bread with or without fructooligosaccharide (a type of dietary fiber) over an 8-week period. Subjects were evaluated regarding their ability to metabolize daidzein to equol.

DETAILED DESCRIPTION:
Soy beans are rich in isoflavones, such as genistein and daidzein, which exhibit estrogenic activity. While the cardiovascular benefits of isoflavones in soy have been recognized, the effects on bone metabolism are less well known. The National Aeronautics and Space Administration expressed an interest in the effects of soy on bone loss and a former NASA scientist developed a soy product, soy bread, which may be more palatable for most Americans than currently available soy foods. A two-treatment two-period crossover trial was conducted to assess the effects of soy bread consumption on deoxypyridinoline, N-telopeptides, bone-specific alkaline phosphatase, osteocalcin, calcium, leptin, insulin-like growth factor-1, luteinizing hormone, follicle-stimulating hormone, testosterone, cholesterol (total, HDL, LDL), triglycerides, apolipoprotein AI, apolipoprotein B, C-reactive protein, and glycosylated hemoglobin. The crossover trial was conducted in subjects identified as having the ability to metabolize daidzein to equol. The treatment was 3 servings of soy bread daily over a 12-week period. The control period included 3 servings of a placebo wheat bread over a 12-week period. For subjects who did not metabolize daidzein to equol at baseline, a pretest-posttest trial of soy bread consumption over an 8-week period was conducted to examine whether 3 servings/day of soy bread increased urinary equol concentrations and whether the addition of fructooligosaccharide enhanced this excretion.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women and men who were 50 years of age or older.

Exclusion Criteria:

* Allergy to soy, wheat, and/or nuts. Use of hormone replacement therapy within the past 6 months. Diagnosis of osteoporosis or use of bone loss medications. Use of drugs within the past 3 months which increase the risk of osteoporosis. End-stage renal disease or other nephropathies. Chemotherapy within the past 6 months. Active gastrointestinal disorders. Diagnosis of thyroid disorder. Use of cholesterol-lowering medications within the past month. Vitamin, mineral, protein, and/or calorie deficiency. Alcoholism, acute or chronic hepatitis, cirrhosis. Use of systemic antibiotics within the past 6 months. Currently under dietary restrictions that would conflict with the intervention. Anticipated mental or physical incapability of adhering to the dietary protocol during the time period of the study (e.g. expected travel).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
deoxypyridinoline | 12 weeks
  Urinary deoxypyridinoline

SECONDARY OUTCOMES:
N-telopeptides, bone-specific alkaline phosphatase, osteocalcin, cholesterol, triglycerides, apolipoproteins, C-reactive protein, HbA1c | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary A.M. Rogers, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States